CLINICAL TRIAL: NCT03881215
Title: Platelet Rich Plasma Following Hysteroscopic Adhesolysis: A Randomized Clinical Trial
Brief Title: Platelet Rich Plasma Following Hysteroscopic Adhesolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AS1811
Record Dates: First submitted 2019-03-16; First posted 2019-03-19 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Intra-uterine Adhesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma (Experimental): PRP
  Interventions: Procedure: Platelet Rich Plasma; Procedure: intra-uterine balloon
- intra-uterine balloon (Active Comparator)
  Interventions: Procedure: intra-uterine balloon

INTERVENTIONS:
Procedure: Platelet Rich Plasma — Platelet Rich Plasma
  Arms: Platelet Rich Plasma
Procedure: intra-uterine balloon — intra-uterine balloon

SUMMARY:
Platelet Rich Plasma Following Hysteroscopic Adhesolysis: A Randomized Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years
* Grade III intra-uterine adhesions

Exclusion Criteria:

* Age < 18 or > 40 years.
* Hb < 11 g/dL, platelets < 150.000/mm3.
* Patient taking anticoagulant.
* Patient taking NSAID in the 10 days before procedure.
* Any significant comorbidity or psychiatric disorder that would compromise patient's consent.
* Active cervical or uterine infection.
* Undiagnosed genital bleeding.
* pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adhesion recurrence | 3 months
  recurrence of severe intra-uterine adhesions

SECONDARY OUTCOMES:
Days of menses | 3 months
  Number of days of menstrual cycle following operation
Amount of menses | 3 months
  Number of sanitary pads changed during each menstrual cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No